CLINICAL TRIAL: NCT03210207
Title: Laparoscopic Gastric Plication: 5 Years of Follow-up in Mexican Patients
Brief Title: Gastric Plication in Mexican Patients
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandro Gonzalez-Ojeda, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: gastroplicature-2017
Record Dates: First submitted 2017-06-27; First posted 2017-07-06 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Bariatric Surgery Candidate; Weight Loss; Obesity, Morbid
MeSH Terms: conditions — Weight Loss; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GASTROPLICATURE: The procedure begins with division of the greater curve vessels from 4 to 5 cm proximal to the pylorus to the angle of His. Either ultrasonic energy or bipolar cautery is appropriate for this step.
  The greater curvature of the stomach is separated from the greater omentum using a harmonic scalpel starting approximately 3cm from the pylorus and ending at or near the angle of His. As needed, adhesions to the posterior surface of the stomach may be transected.
  At least two rows of at least five continuous stitches will be placed laparoscopically about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum
  Interventions: Procedure: GASTROPLICATURE

INTERVENTIONS:
Procedure: GASTROPLICATURE — All procedures were performed by a single surgeon. All patients underwent 2-row gastric plication. Dissection was started at the greater curvature of the stomach in contact to the gastric wall from prepyloric area to 2-cm proximal to the Hiss angle preserving the anatomy of Hiss angle. All vessels along the greater curvature were separated using LigaSure (Covidien, Mansfield, MA, USA). The greater curvature (from the perimeter) was invaginated using 2 rows of 00 prolene or 00 nylon sutures. Two layers of plication were performed with continuous sutures with 1 surgical sting in all patients to prevent any displacement of inverted folds such as eversion outside or intussusception into esophagus or pylorus. All sutures were extramucusal to avoid their absorption by gastric acid. Finally, a tube shaped stomach was achieved in which the greater curvature was inverted in to the stomach.

SUMMARY:
Between January and December 2012, a total of 40 patients underwent GLP. The study will assess subject excess weight loss (%EWL) following the study procedure at 3, 6, 12, 36 and 60 months.

DETAILED DESCRIPTION:
The patient characteristics extracted from the medical records included age and gender. A detailed height and weight history was collected to reflect BMI, excess weight, %EWL, and %BMI before LGP and after 3, 6, 12, 36 and 60 months.

The institutional review board approved the present study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to give consent and comply with evaluation and treatment schedule for female patients, this includes agreement to use a reliable (per investigator) form of birth control for the duration of the trial)
* 18 to 50 years
* Subject meets ASMBS and NIH criteria: (consensus.nih.gov)
* BMI ³ 40 kg/m2 and £ 50 kg/m2; or, BMI 35-40 kg/m2 with one or more significant co-morbid medical conditions which are generally expected to be improved, reversed, or resolved by weight loss, including:
* Hyperlipidemia
* Mild obstructive sleep apnea (per Investigator discretion)
* Hypertension
* Osteoarthritis of the hip or knee per investigational site's criteria for which the subject is being treated;
* ASA Class I - III;
* Agree to refrain from any type of weight-loss drug (prescription or OTC) or elective procedure that would affect body weight for the duration of the trial;
* HbA1C < 11%; and
* For subjects who have Type 2 diabetes, medication regimen is no more complex (2 oral medications) than oral metformin plus one oral sulfonylurea plus once daily insulin injection.

Exclusion Criteria:

* Documented history of drug and/or alcohol abuse within two (2) years of the Screening Visit;
* Previous malabsorptive or restrictive procedures performed for the treatment of obesity;
* Scheduled concurrent surgical procedure, with the exception of SOC liver biopsy;
* Women of childbearing potential who are pregnant or lactating at the time of screening or at the time of surgery;
* Psychiatric disorders that may affect compliance with the clinical trial, including dementia, active psychosis, severe depression requiring > 2 medications, or history of suicide attempts;
* Participation in any other investigational device or drug study (non-survey based trial; long-term enrollment in such studies as requiring periodic laboratory tests, etc., would be allowed) within 12 weeks of enrollment
* Any condition which precludes compliance with the study, including:
* Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis that have been active within the past 10 years;
* Congenital or acquired anomalies of the GI tract, including atresias or stenosis;
* Severe cardiopulmonary disease or other serious organic disease that makes the subject a high-risk surgical candidate;
* Uncontrolled hypertension;
* Portal hypertension;
* Chronic or acute upper gastrointestinal bleeding conditions (e.g., gastric or esophageal varices);
* Cirrhosis;
* Congenital or acquired intestinal telangiectasia;
* Esophageal or gastric disorders including moderate severe preoperative reflux, dysmotility, or Barrett's esophagus;
* Presence of hiatal hernia greater than 2cm in length, with the exception of a small sliding hiatal hernia previously undiagnosed and discovered during the surgical procedure;
* Prior surgery of the foregut including hiatal hernia repair or prior gastric surgery;
* Known history of clotting disorders, hemoglobinopathies, and hemolytic disorders, including pulmonary embolus and Deep Vein Thrombosis;
* Pancreatitis;
* Gallstones (confirmed via ultrasound);
* Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
* Use of thiazolidinediones ("glitazones"), or Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study;
* History or presence of pre-existing autoimmune connective tissue disease;
* Use of prescription or over the counter weight reduction medications or supplements within thirty days of the Screening Visit or the duration of study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mexican patients who underwent Gastroplicature
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
excess weight loss (%EWL) | 3 postoperative months
weight loss | 3 postoperative months
BMI loss | 3 postoperative months
excess of BMI loss (%BMI) | 3 postoperative months
%EWL | 6 postoperative months
%EWL | 12 postoperative months
%EWL | 36 postoperative months
%EWL | 60 postoperative months
weight loss | 6 postoperative months
weight loss | 12 postoperative months
weight loss | 36 postoperative months
weight loss | 60 postoperative months
BMI loss | 6 postoperative months
BMI loss | 12 postoperative months
BMI loss | 36 postoperative months
BMI loss | 60 postoperative months
%BMI | 6 postoperative months
%BMI | 12 postoperative months
%BMI | 36 postoperative months
%BMI | 60 postoperative months

IPD SHARING:
Plan to Share IPD: No